CLINICAL TRIAL: NCT03187470
Title: The Impact of Multipole Pacing (MPP) on Left Ventricular Dyssynchrony in Patients With Cardiac Resynchronization Therapy (CRT) - a Real-Time Three Dimensional Echocardiography Approach
Brief Title: Left Ventricular Dyssynchrony in Multipole Pacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adnan Kastrati, MD (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor-Investigator, Adnan Kastrati, MD, Prof. Dr. Adnan Kastrati, Deutsches Herzzentrum Muenchen
Organization: Deutsches Herzzentrum Muenchen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: GER-EP-016
Record Dates: First submitted 2017-04-10; First posted 2017-06-15 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Different programming of a CRT defibrillator — Different programming of a CRT defibrillator using pacing modalities of a quadripolar left ventricular lead

SUMMARY:
Left ventricular dyssynchrony will be assessed by echocardiography using different programming of an implantable cardioverter defibrillator.

DETAILED DESCRIPTION:
Left ventricular dyssynchrony will be assessed by echocardiography using different programming of an implantable cardioverter defibrillator using a quadripolar left ventricular lead.

ELIGIBILITY:
Inclusion Criteria:

* Indication for the implantation of a defibrillator with cardiac resynchronisation therapy

Exclusion Criteria:

* Cardiac surgery, acute coronary syndrome / myocardial infarction, percutaneous coronary intervention within the past 4 weeks
* Indication for coronary artery revascularisation
* Atrial fibrillation with insufficient rate control
* ASA (American Society of Anesthesiologists) class V or cardiogenic shock
* age <18 years, pregnancy, tutelage
* inability to understand the patient consent for or study refusal
* anticipated insufficient echocardiographic image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Left ventricular dyssynchrony | 15 minutes
  Left ventricular dyssynchrony

SECONDARY OUTCOMES:
left ventricular ejection fraction | 15 minutes
  left ventricular ejection fraction

CONTACTS AND LOCATIONS:
Overall Officials: Severin Weigand, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum München, München, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weigand S, Karl M, Brkic A, Lennerz C, Grebmer C, Blazek P, Kornmayer M, Schaarschmidt C, Wesemann L, Reents T, Hessling G, Deisenhofer I, Kolb C. The impact of multipole pacing on left ventricular function in patients with cardiac resynchronization therapy - A real-time three-dimensional echocardiography approach. Int J Cardiol. 2018 Dec 1;272:238-243. doi: 10.1016/j.ijcard.2018.08.033. Epub 2018 Aug 15. PMID 30121181